CLINICAL TRIAL: NCT00994773
Title: A Pilot Trial of Simvastatin Alone and Added to Tenofovir or Entecavir for the Treatment of Chronic Hepatitis B
Brief Title: Simvastatin for the Treatment of Chronic Hepatitis B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bader, Ted, M.D. (Individual)
Responsible Party: Principal Investigator, Ted Bader, MD, Director of Liver Diseases, OUHSC/VAMC, Bader, Ted, M.D.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBV 14934; Simvastatin against HepB
Record Dates: First submitted 2009-10-10; First posted 2009-10-14 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; simvastatin; HBV DNA
MeSH Terms: conditions — Hepatitis B | interventions — Simvastatin; Tenofovir; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Simvastatin (Experimental): Simvastatin orally
  Interventions: Drug: Simvastatin
- Simvastatin and tenofovir (Experimental): Simvastatin combined with tenofovir
  Interventions: Drug: Simvastatin; Drug: Tenofovir
- Simvastatin and entecavir (Experimental): Simvastatin combined with entecavir
  Interventions: Drug: Simvastatin; Drug: Entecavir

INTERVENTIONS:
Drug: Simvastatin — daily doses for 14 days
  Other Names: Zocor
Drug: Tenofovir
  Arms: Simvastatin and tenofovir
Drug: Entecavir — Entecavir
  Arms: Simvastatin and entecavir

SUMMARY:
The investigators have shown robust in vitro anti-hepatitis B activity of simvastatin alone and synergistic activity with all four FDA-approved anti-hepatitis B oral drugs tested. The investigators propose phase 1 studies in 48 chronic hepatitis B human carriers who have never been treated before. Doses of drugs will remain at or below FDA-approved dosage levels for cholesterol lowering (simvastatin) or hepatitis B (tenofovir or entecavir). Arm 1 will have simvastatin monotherapy only. Arm 2 will combine simvastatin with tenofovir. Arm 3 will combine simvastatin with entecavir. For maximum safety, the 3 arms and the dose groups in each arm will be filled consecutively and not concurrently. The definition of efficacy for simvastatin alone will be a 1 log drop of hepatitis B virus in 14 days. Efficacy for combination of drugs will require a 2 log drop of hepatitis B virus in 14 days. Numerous safety tests and stop rules are noted in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Hepatitis B positive by HBV DNA within 180 days.
2. Ages 18-70.
3. Men and non-pregnant women eligible.
4. Veteran's eligibility or appropriate health insurance.

Exclusion Criteria:

1. Use of any anti-HBV medicine within 30 days.
2. Decompensated cirrhosis as evidenced by esophageal varices, ascites, or encephalopathy. (grade 1 varices without history of bleeding will be allowed, if patient meets Child's-Pugh functional classification grade A).
3. A positive urine test for marijuana or alcohol within 2 months of screening.(Allowed to repeat tests on different days, if positive first time in order to become eligible for study.
4. Severe cardiovascular disease (ejection fraction <20%)* or uncontrolled angina.
5. Severe pulmonary disease (FEV1 < 1.0).
6. Chronic renal insufficiency (creatinine clearance <50 ml/min.
7. HIV positive patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Reduction of HBV DNA by one log. | 14 days
  Simvastatin will be given in doses of 5,10,20,and 40mg per day

SECONDARY OUTCOMES:
Alanine aminotransferase (ALT) reduction | 14 days
  ALT changes will be noted

CONTACTS AND LOCATIONS:
Overall Officials: Teddy Bader, M.D., Principal Investigator — University of Oklahoma
Locations (1):
- VA Medical Center, Oklahoma City, Oklahoma, United States